CLINICAL TRIAL: NCT06505356
Title: Characterization of Microbiological and Genetic Features in Prostate Cancer Patients and Their Associations with Disease Stage and Clinical Presentation
Brief Title: Characterization of Microbiological and Genetic Features in Prostate Cancer and Their Association with Disease Stage
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Edgaras Burzinskis (Other)
Responsible Party: Sponsor-Investigator, Edgaras Burzinskis, Principal Investigator, Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Nr. BE-2-10
Record Dates: First submitted 2024-06-04; First posted 2024-07-17 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer; Prostate Inflammation
MeSH Terms: conditions — Prostatic Neoplasms; Prostatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with diagnosed prostate cancer after TRUS prostate biopsy (Experimental): Prostate Biopsy Procedure (TRUS-guided): Preparation: Explain procedure, obtain consent. Administer antibiotics, discontinue blood thinners. No bowel prep needed. Procedure: Position: Patient lies on side or in lithotomy position. Anesthesia: Apply local anesthetic. Insert ultrasound probe into rectum to visualize prostate. Guide needle into prostate using ultrasound. Take 10-12 tissue samples. Post-procedure: Monitor for complications. Continue antibiotics, drink fluids, avoid strenuous activity. Side Effects: Minor blood in urine, semen, or rectum, resolving in days to weeks. Follow-up: Discuss results within a week. Expected result: confirmation of prostate cancer.
  Interventions: Procedure: Prostate biopsy
- Patients without a prostate cancer diagnosis after TRUS prostate biopsy (Experimental): Experimental: Patients without a prostate cancer diagnosis after TRUS biopsy. Prostate Biopsy (TRUS-guided). Preparation: Explain procedure, benefits, and risks; obtain consent. Administer antibiotics; discontinue blood thinners. No bowel prep. Procedure: Patient lies on their side or in lithotomy position. Apply local anesthetic. Insert lubricated ultrasound probe into rectum. Guide thin needle into prostate using ultrasound. Take 10-12 tissue samples. Post-procedure: Monitor for complications. Continue antibiotics, drink fluids, avoid strenuous activity, monitor for complications. Minor blood in urine, semen, or rectum may occur, resolving in days to weeks. Follow-up: Discuss biopsy results within a week. Expected result: Absence of prostate cancer.
  Interventions: Procedure: Prostate biopsy

INTERVENTIONS:
Procedure: Prostate biopsy — Transrectal prostate biopsy

SUMMARY:
1. Identify the local inflammatory response in prostate tissue and the systemic response in the blood of patients with prostate cancer, depending on the stage of the disease, and evaluate their prognostic value.
2. Identify the spectrum of microorganisms and antibiotic resistance in patients with prostate cancer prior to prostate biopsy, and assess the risk of complications when using Ciprofloxacin and Fosfomycin.
3. Determine the significance of GAS5, JAZF1, and CTBP2 gene polymorphisms in the development of prostate cancer.
4. Evaluate the association of a specific gene polymorphism with the clinical course of the disease in patients with prostate cancer.

DETAILED DESCRIPTION:
Goal 1: Identify Local Inflammatory Response in Prostate Tissue and Systemic Response in the Blood of Patients with Prostate Cancer Depending on the Stage of the Disease and Evaluate Their Prognostic Value

Objective: To investigate and characterize both local and systemic inflammatory responses in prostate cancer patients at various disease stages.

Approach:

* Local Inflammatory Response: Examine prostate tissue samples to identify markers and levels of inflammation. This involves histological analysis and possibly molecular assays (e.g., PCR, immunohistochemistry).
* Systemic Inflammatory Response: Measure inflammatory markers in the blood, such as C-reactive protein (CRP), interleukins (e.g., IL-6), and other cytokines.
* Disease Staging: Correlate these inflammatory responses with the stage of prostate cancer (e.g., localized, advanced, metastatic) to understand the progression of the disease.
* Prognostic Value: Analyze the data to determine if these inflammatory markers can predict disease progression, response to treatment, and overall prognosis.

Expected Outcome: Establish a comprehensive profile of inflammatory responses associated with different stages of prostate cancer and identify potential prognostic biomarkers.

Goal 2: Identify the Spectrum of Microorganisms and Antibiotic Resistance in Patients with Prostate Cancer Prior to Prostate Biopsy and Assess the Risk of Complications When Using Ciprofloxacin and Fosfomycin

Objective: To profile the microbial flora and antibiotic resistance in prostate cancer patients before biopsy, and evaluate the safety and efficacy of Ciprofloxacin and Fosfomycin.

Approach:

* Microbial Spectrum: Collect and analyze urine, prostatic fluid, and other relevant samples to identify bacterial species present using culture methods and molecular techniques.
* Antibiotic Resistance: Test the identified microorganisms for resistance to common antibiotics, focusing on Ciprofloxacin and Fosfomycin.
* Risk Assessment: Review patient outcomes post-biopsy to assess the incidence of complications such as infection and adverse reactions, particularly in relation to the use of the studied antibiotics.
* Data Analysis: Correlate microbial profiles and resistance patterns with clinical outcomes to determine the risk factors for complications.

Expected Outcome: Develop guidelines for antibiotic use in prostate biopsy procedures based on microbial and resistance profiles to minimize the risk of complications.

Goal 3: Determine the Significance of GAS5, JAZF1, and CTBP2 Gene Polymorphism in the Development of Prostate Cancer

Objective: To investigate the role of specific gene polymorphisms (GAS5, JAZF1, and CTBP2) in the susceptibility to and development of prostate cancer.

Approach:

* Genetic Analysis: Collect DNA samples from prostate cancer patients and a control group. Perform genotyping to identify polymorphisms in the GAS5, JAZF1, and CTBP2 genes.
* Association Studies: Conduct statistical analyses to compare the frequency of these polymorphisms in patients versus controls. Assess their correlation with the presence and severity of prostate cancer.
* Functional Studies: Where possible, explore the biological impact of these polymorphisms on gene expression and function, potentially through in vitro or in vivo models.

Expected Outcome: Identify genetic markers that contribute to prostate cancer risk, enhancing understanding of disease mechanisms and potential targets for intervention.

Goal 4: Evaluate the Associations of One Gene Polymorphism with the Clinical Course of Disease in Patients with Prostate Cancer

Objective: To determine how a specific gene polymorphism influences the clinical trajectory of prostate cancer.

Approach:

* Polymorphism Selection: Choose a gene polymorphism of interest, potentially based on findings from previous research or Goals 1-3.
* Clinical Data Collection: Gather comprehensive clinical data from prostate cancer patients, including disease stage, progression, treatment response, and outcomes.
* Genotype-Phenotype Correlation: Perform genetic testing to identify the presence of the polymorphism in these patients. Correlate the genetic data with clinical parameters to assess associations.
* Statistical Analysis: Use appropriate statistical methods to determine the significance of the associations between the polymorphism and various clinical aspects of prostate cancer.

Expected Outcome: Gain insights into how genetic variations can affect the progression and treatment response in prostate cancer, potentially guiding personalized treatment approaches.

Prostate Cancer and Biopsy Related Acronyms:

1. TRUS: Transrectal Ultrasound

   * A medical imaging technique used to visualize the prostate gland and guide the biopsy needle.
2. PSA: Prostate-Specific Antigen

   * A protein produced by the prostate gland, elevated levels of which can indicate prostate cancer.
3. Gleason Score:

   * A grading system used to determine the aggressiveness of prostate cancer based on the microscopic appearance of prostate tissue.

Genetic and Molecular Biology Acronyms:

1. GAS5: Growth Arrest Specific 5

   * A long non-coding RNA involved in regulating cell growth and apoptosis, often studied in cancer research.
2. JAZF1: JAZF Zinc Finger 1

   * A gene associated with various cellular processes, including transcriptional regulation and potentially linked to cancer.
3. CTBP2: C-terminal Binding Protein 2

   * A protein that functions as a transcriptional co-repressor, playing a role in gene expression regulation and cancer.
4. PCR: Polymerase Chain Reaction

   * A laboratory technique used to amplify DNA sequences, making it easier to study genetic material in detail.
5. NGS: Next-Generation Sequencing

   * Advanced sequencing technologies that allow for rapid and detailed sequencing of large amounts of DNA.

Inflammatory Markers:

1. 6Ckine (CCL21): Chemokine (C-C motif) ligand 21

   * A cytokine involved in the immune response and potentially linked to inflammation in cancer.
2. Eotaxin (CCL11): Chemokine (C-C motif) ligand 11

   * A chemokine that attracts eosinophils and is associated with allergic responses and inflammation.
3. Fractalkine (CX3CL1): Chemokine (C-X3-C motif) ligand 1

   * A chemokine involved in immune cell migration and adhesion, playing a role in inflammation and cancer.
4. IFN gamma: Interferon gamma

   * A cytokine critical for innate and adaptive immunity against viral and intracellular bacterial infections and for tumor control.
5. IL-2: Interleukin 2

   * A cytokine that promotes the growth and differentiation of T cells, important in the immune response.
6. IL-6: Interleukin 6

   * A cytokine involved in inflammation and infection responses, also linked to cancer progression.
7. IL-8 (CXCL8): Interleukin 8

   * A chemokine that attracts neutrophils and is involved in the inflammatory response.
8. IL-10: Interleukin 10

   * A cytokine with anti-inflammatory properties, regulating immune responses.
9. IL-18: Interleukin 18

   * A cytokine that induces interferon gamma production, playing a role in inflammation and immune responses.
10. MIP-3 beta (CCL19): Macrophage Inflammatory Protein 3 beta

    * A chemokine involved in immune cell trafficking and inflammatory responses.
11. PDGF-BB: Platelet-Derived Growth Factor BB

    * A growth factor involved in blood vessel formation and the growth of various cell types.
12. TNF alpha: Tumor Necrosis Factor alpha

    * A cytokine involved in systemic inflammation and is part of the immune system's response to cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Male patients aged 18 years and older.
2. Diagnosis: Patients who are suspected of having prostate cancer based on clinical data and standard diagnostic protocols.
3. Disease Stage: Patients at any stage of suspected prostate cancer (localized, locally advanced, or metastatic).
4. Consent: Ability and willingness to provide written informed consent.
5. Clinical Data Availability: Availability of comprehensive clinical data.
6. Sample Provision: Willingness to provide blood and/or tissue samples for genetic and inflammatory marker analysis.

Exclusion Criteria:

1. Prior Treatment: Patients who have undergone any prior prostate cancer treatments such as surgery, radiation therapy, or systemic therapies (e.g., hormone therapy, chemotherapy).
2. Other Malignancies: Presence of other concurrent malignancies, except for adequately treated basal cell or squamous cell skin cancer.
3. Severe Comorbidities: Patients with severe or uncontrolled comorbid conditions that could interfere with study participation or data interpretation (e.g., severe cardiovascular, pulmonary, hepatic, or renal diseases).
4. Infection: Active infections or other severe medical conditions that could compromise patient safety or study integrity.
5. Non-compliance: Inability to comply with study procedures, follow-up requirements, or any condition that, in the investigator's opinion, could interfere with study participation.
6. Medication Use: Use of medications that could interfere with the study results, such as immunosuppressive drugs.

Additional Considerations:

* Screening: All potential participants will undergo a screening process to verify eligibility criteria.
* Confidentiality: Ensure all patient data is handled in accordance with privacy regulations and ethical guidelines.
* Follow-Up: Participants should be willing to attend regular follow-up visits for ongoing data collection and monitoring of disease progression and treatment response.

By setting these criteria, the study aims to create a well-defined patient cohort for evaluating the relationship between genetic and inflammatory markers and prostate cancer aggressiveness.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study includes male participants as defined by their self-identified gender. This approach ensures inclusivity and respects the gender identity of all participants. Participants must have a prostate, which is an organ typically found in males.
Enrollment: 400 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Inflammatory markers' effect on prostate cancer aggressiveness | 2 weeks
  Aim: Assess if selected inflammatory markers are linked to prostate cancer aggressiveness by measuring their concentrations and analyzing correlations with disease severity.
  Markers:
  6Ckine (CCL21) Eotaxin (CCL11) Fractalkine (CX3CL1) IFN gamma IL-2 IL-6 IL-8 (CXCL8) IL-10 IL-18 MIP-3 beta (CCL19) PDGF-BB TNF alpha
  Objectives:
  1. Measure marker levels in blood samples.
  2. Investigate links between marker levels and cancer aggressiveness.
  3. Use Gleason score, seminal vesicles invasion, and lymph nodes invasion.
  Outcomes:
  Identify markers linked to aggressiveness. Develop prognostic tools or therapies. Categorize patients by risk. This study aims to understand inflammation's role in prostate cancer and identify biomarkers for predicting aggressiveness.
Genetic polymorphism markers' effect on prostate cancer aggressiveness | 2 weeks
  Genetic Polymorphism Markers' Effect on Prostate Cancer Aggressiveness
  Objectives:
  1. Examine GAS5, JAZF1, CTBP2 polymorphisms and their variations in patients.
  2. Measure polymorphism levels and their relationship with cancer aggressiveness.
  3. Correlate polymorphisms with Gleason score, seminal vesicles invasion, and lymph nodes invasion.
  Expected Outcomes:
  * Identify markers linked to aggressiveness.
  * Provide insights for genetic tests.
  * Understand molecular mechanisms and develop therapies. This study clarifies the role of genetic polymorphisms in prostate cancer aggressiveness, aiding prognosis and treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided